CLINICAL TRIAL: NCT03119584
Title: Efficacy of Linaclotide in Type II Diabetics With Chronic Constipation: A Randomized, Double-Blind, Placebo-Controlled, Cross-Over Trial
Brief Title: Efficacy of Linaclotide in Type II Diabetics With Chronic Constipation
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Irene Sarosiek, Professor of Medicine, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: E15025
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Chronic Constipation; Diabete Mellitus
Keywords: chronic constipation; diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1)28days of linaclotide or placebo (Active Comparator): patient will be randomized and allocated to one of the treatment arms using computerized generated simple random number in a double-blinded fashion for 28 days of therapy with the study drug, linaclotide or placebo. Patients, and trial personnel involve (other than biostatistician) in this study will not be aware of the group assignments. Patients, treatment providers and staffs will be kept blinded in this study.
  Interventions: Drug: linaclotide or placebo
- 2)28days of linaclotide or placebo (Active Comparator): patient will be randomized and allocated to one of the treatment arms using computerized generated simple random number in a double-blinded fashion for 28 days of therapy with the study drug, linaclotide or placebo. Patients, and trial personnel involve (other than biostatistician) in this study will not be aware of the group assignments. Patients, treatment providers and staffs will be kept blinded in this study.
  Interventions: Drug: linaclotide or placebo

INTERVENTIONS:
Drug: linaclotide or placebo
  Other Names: Linzess

SUMMARY:
Study includes 5 visits, when all basic clinical information, vital signs, symptoms, and side effects are going to be assessed at each appointment.

Patients are going to be assigned by the computer, to receive an active or non-active drug for 14 days in a first phase. The order will be change during the second phase. The 2 weeks break without our medication will separate these phases. A very close observation regarding safety of our subjects will be implemented by study personnel and clinical investigators.

DETAILED DESCRIPTION:
The symptoms of chronic constipation are defined as infrequent bowel movements, hard stool, straining during defecation, bloating, abdominal discomfort, and sensation of incomplete evacuation.

Constipation has been reported as a common complication of diabetic neuropathy. A new medication, called linaclotide, was studied on many patients, and it is approved to be on a market for constipated patients. Unfortunately diabetics were not included in these previous studies; hence we designed the project which is going to address the possible benefit of this drug in diabetic population.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetics.
* Functional Constipation defined by Rome III criteria are as follows: a. At least a 6 months history of constipation.

  b. Less than three spontaneous bowel movements (SBMs) per week. c. At least 25% of stools are lumpy or hard stools as it is described in Bristol Stool Form Scale (BSFS) less than score of 6.

  d. Sensation of incomplete evacuation following at least 25% of bowel movements.

  e. Straining on at least 25% of defecations. f. Sensation of anorectal obstruction/blockage for at least 25% of defecations.

Note: The above criteria are only applicable to spontaneous bowel movements. Patients who have no spontaneous bowel movements (bowel movements are preceded by laxative intake) are considered constipated and are eligible for this study.

* For patients' ≥ 50 years of age, normal colonic anatomy as documented by colonoscopy or double-contrast barium enema, performed within the previous 5 years, based on the American Gastroenterological Association guidelines.
* Patients with confirm diagnosis of Diabetic Autonomic Neuropathy based on results of ANX 3.0, real-time ANS monitoring system will be included in this investigation.
* Patients diagnosed with diabetic peripheral neuropathy and/or symptoms of functional gastroduodenal disorders, such as GERD and functional dyspepsia may participate in a study.

Exclusion Criteria:

* Pregnancy or lactation
* Subjects unwilling to practice adequate contraception throughout the period of screening through 14 days after study termination.
* Loose or watery stools reported in the absence of laxatives for >25% of BMs during the screening period by using Bristol Stool Form Scale (BSFS).
* Use of laxatives 3 days immediately prior to randomization (except fiber or bulking agents) and chronic laxative use during the trial.
* Patients diagnosed with severe, drug refractory gastroparesis (persistent daily vomiting), currently receiving parenteral feeding (N-G, J-G-Tubes), having history of frequent hospitalizations, or being implanted with gastric neurostimulation system.
* Use of any of the following drugs within 3 days prior randomization and during the trial: a. Prokinetic agents (domperidone, metoclopramide, erythromycin).

  b. Medication containing opiates. c. Anti-spasmodic (e.g. Atropine, hyoscamine, scopolamine, glycopyrrolate).
* Hemoglobin A1c>8.2
* Use of illegal drugs.
* Regular consumption of more than 2 drinks of alcohol per day
* Chronic, more than 3/week use of NSAIDs.
* Patients with prolonged straining/push during BMs suggesting severe pelvic floor dysfunction.
* History or current diagnosis of diverticulitis and severe hemorrhoids.
* History of gastric resections, partial colon resection, history of rectocele.
* Existence of any major medical condition such as malignancy, severe renal and liver diseases, which in the decision of PI should be excluded from participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in frequency of bowel movements | Up to 10 weeks
  The primary outcome measure will indicate improvement in frequency of bowel movements (BMs) or not in a mean of available and recordered spontaneous BM (SBMs) over the 28 day treatment period compared to 28 days of placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Sarosiek, MD, Principal Investigator — Texas Tech University Health Sciences Center- El Paso, Texas
Locations (1):
- Texas Tech University Health Sciences Center, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No